CLINICAL TRIAL: NCT06707506
Title: CT-Derived Metabolic Parameters as Predictors of Post-Operative Atrial Fibrillation Following Minimally Invasive Mitral Valve Surgery: The MiniMitral AF Study
Brief Title: Atrial Fibrillation Risk After Miniinvasive Mitral Valve Repair
Status: Completed | Type: Observational
Sponsor: Nemocnice AGEL Trinec-Podlesi a.s. (Other)
Responsible Party: Principal Investigator, Matej Pekar, MD, PhD, Matej Pekar, MD, PhD, Nemocnice AGEL Trinec-Podlesi a.s.
Other Study IDs: EK 65/24
Record Dates: First submitted 2024-11-24; First posted 2024-11-27 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Mitral Regurgitation; Computed Tomography; Atrial Fibrillation
Keywords: Post-operative Atrial Fibrillation; Body Composition; Computed Tomography; Mitral Valve Surgery; Metabolic Risk Factors
MeSH Terms: conditions — Mitral Valve Insufficiency; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This retrospective cohort study investigates how CT-derived tissue quality parameters, serving as markers of metabolic status, predict post-operative atrial fibrillation risk in patients undergoing minimally invasive mitral valve surgery. The study leverages established associations between adipose tissue characteristics and metabolic dysfunction to explore their potential role in post-surgical arrhythmogenesis.

DETAILED DESCRIPTION:
Scientific Background and Rationale Post-operative atrial fibrillation (POAF) affects up to 30% of patients following cardiac surgery and significantly impacts outcomes. While traditional risk factors are well-documented, the role of underlying metabolic dysfunction in arrhythmogenesis remains poorly understood. Recent evidence suggests that tissue-specific metabolic alterations, particularly in adipose tissue distribution and quality, may provide crucial insights into arrhythmic risk. CT-derived tissue quality parameters (measured in Hounsfield Units) have been validated as markers of metabolic status, with studies demonstrating associations between adipose tissue density and inflammatory states. This study aims to investigate whether these metabolic markers can predict POAF risk in the specific context of mitral valve surgery, potentially informing risk stratification and preventive strategies.

Primary Objective To determine whether CT-derived tissue quality parameters (adipose tissue density, muscle density) independently predict post-operative atrial fibrillation risk following minimally invasive mitral valve surgery.

Study Design

Observational Model: Retrospective Cohort Setting: Single-center study at Complex Cardiovascular Center, Hospital AGEL Trinec-Podlesi Time Frame: January 2014 - November 2023 Follow-up: Through August 1, 2024

Primary Outcome Measure Post-operative Atrial Fibrillation [Time Frame: Up to 30 days post-surgery]

Defined as new-onset AF lasting more than 48 hours or requiring intervention Measured through continuous cardiac monitoring Analyzed separately for patients with and without preoperative AF history

Secondary Outcome Measures

Overall Survival [Through August 1, 2024]

Perioperative Complications:

Blood product utilization Duration of mechanical ventilation ICU length of stay Total hospital length of stay

Key Study Groups

AF-Naïve Group (n=56):

No previous AF history Primary prevention cohort

AF-History Group (n=48):

Preexisting AF with concurrent Maze procedure Secondary prevention cohort

CT Analysis Methods

Automated segmentation at L3 vertebral level

Parameters measured:

Muscle density (HU) Intramuscular adipose tissue density (IMAT HU) Visceral adipose tissue density (VAT HU) Subcutaneous adipose tissue density (SAT HU) Skeletal muscle index (SMI)

Statistical Analysis Plan

Primary analysis: Logistic regression for POAF prediction Interaction analysis between tissue parameters and AF history Adjustment for age, gender, and traditional risk factors Separate models for AF-naïve and AF-history groups

Eligibility Criteria

Inclusion Criteria:

Age ≥ 18 years Undergoing minimally invasive mitral valve surgery Preoperative CT scan available Surgery between January 2014 and November 2023

Exclusion Criteria:

Incomplete clinical data Poor quality CT images Previous cardiac surgery

Sample Size 114 total participants (104 included in primary analysis) Study Status

Completed enrollment Final follow-up: August 1, 2024 Ethics Committee Approval: EK 65/24

Principal Investigators

Matej Pekar, MD David Vician, MD Complex Cardiovascular Center, Hospital AGEL Trinec-Podlesi

Funding Sources

MUNI/A/1547/2023 MUNI/A/1555/2023 Ministry of Education, Youth, and Sports of the Czech Republic

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Undergoing minimally invasive mitral valve surgery
* Preoperative CT scan available
* Surgery between January 2014 and November 2023

Exclusion Criteria:

* Incomplete clinical data
* Poor quality CT images
* Previous cardiac surgery

Ages: 19 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This single-center retrospective cohort study included 114 consecutive patients who underwent minimally invasive mitral valve surgery between January 2014 and November 2023 at the Complex Cardiovascular Center, Hospital AGEL Trinec-Podlesi.
Sampling Method: Non-Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
postoperative atrial fibrillation development | Through August 1, 2024
  Defined as new-onset AF lasting more than 48 hours or requiring intervention Measured through continuous cardiac monitoring Analyzed separately for patients with and without preoperative AF history

SECONDARY OUTCOMES:
Overall Survival | Through August 1, 2024
  Overall Survival in the cohort
Perioperative Complications | Through August 1, 2024
  Blood product utilization Duration of mechanical ventilation ICU length of stay Total hospital length of stay